CLINICAL TRIAL: NCT02065089
Title: Development of an Electronic Pediatric Inflammatory Bowel Disease Quiz
Brief Title: Development of 'Emma'--a Pediatric IBD Quiz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeanne Tung, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-000584
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Ulcerative Colitis; Crohn's Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- playing the ipad quiz game (Experimental): There will only be one arm--any patient who consents to participate in the intervention (playing the ipad quiz game)
  Interventions: Other: playing the ipad quiz game

INTERVENTIONS:
Other: playing the ipad quiz game — Individualized education to the patient via the quiz game, with optional additional education provided by medical providers.

SUMMARY:
We would like to collaborate and further develop an ipad-based, interactive quiz game 'Emma'; to identify gaps in knowledge of inflammatory bowel disease in pediatric patients. These gaps can be used to improve patient education.

ELIGIBILITY:
Inclusion Criteria:

* Children 10-18 years of age
* Diagnosis of Crohn's disease or ulcerative colitis
* English-speaking
* Established patient of participating institution

Exclusion criteria

* Inability to understand and read English at a grade 5-12 year level, as commensurate to their chronological age
* Research denial by patient or guardian

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Improvement in patient knowledge of inflammatory bowel disease | baseline to 18 months
  The patient will play the ipad quiz game at office visits over time. We will look for improvements in overall knowledge of IBD, as well as subcategories (ex. nutrition, medications, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Tung, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma